CLINICAL TRIAL: NCT02390882
Title: A Multicenter, Randomized, Double-blind, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of HGP0412 and HIP1402 in Patients With Benign Prostatic Hyperplasia
Brief Title: A Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of HGP0412 and HIP1402 in Patients With BPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-VICT-301
Record Dates: First submitted 2015-02-23; First posted 2015-03-18 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Benign Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Tamsulosin placebo (12 weeks)
  Interventions: Drug: Placebo
- Treatment 1 (Experimental): HGP0412 capsule (12 weeks)
  Interventions: Drug: HGP0412 capsule
- Treatment2 (Experimental): HIP1402 capsule (12 weeks)
  Interventions: Drug: HIP1402 capsule

INTERVENTIONS:
Drug: Placebo — Placebo
  Other Names: Tamsulosin Placebo
  Arms: Placebo
Drug: HGP0412 capsule — Tamsulon high dose
  Other Names: Tamsulosin HCl 0.2mg
  Arms: Treatment 1
Drug: HIP1402 capsule — Tamsulon high dose
  Other Names: Tamsulosin HCl 0.4mg
  Arms: Treatment2

SUMMARY:
The main objective of this study is to evaluate efficacy and safety of (Tamsulosin) HGP0412 and HIP1402 in patients with Benign Prostatic Hyperplasia

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, phase 3 clinical trial to evaluate the efficacy and safety of (Tamsulosin) HGP0412 and HIP1402 in patients with benign prostatic hyperplasia

ELIGIBILITY:
Inclusion Criteria:

* age>=45, male, diagnosed on BPH, Total IPSS>=13

Exclusion Criteria:

* Hypersensitivity to investigational products or components
* PSA>=4ng/ml

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Total International Prostate Symptom Score | 12 weeks

SECONDARY OUTCOMES:
Total International Prostate Symptom Score | 4, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lee, MD, Principal Investigator — Hanyang University Guri Hospital
Locations (1):
- Hanyang University Guri Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung JH, Oh CY, Kim JH, Ha US, Kim TH, Lee SH, Han JH, Bae JH, Chang IH, Han DH, Yoo TK, Chung JI, Kim SW, Jung J, Kim YI, Lee SW. Efficacy and safety of tamsulosin 0.4 mg single pills for treatment of Asian patients with symptomatic benign prostatic hyperplasia with lower urinary tract symptoms: a randomized, double-blind, phase 3 trial. Curr Med Res Opin. 2018 Oct;34(10):1793-1801. doi: 10.1080/03007995.2018.1447451. Epub 2018 Apr 12. PMID 29490509